CLINICAL TRIAL: NCT00584519
Title: Control of Metabolic and Cardiovascular Risk in Patients With Schizophrenia and Overweight (CRESSOB)
Brief Title: Control of Metabolic and Cardiovascular Risk in Patients With Schizophrenia and Overweight
Acronym: CRESSOB
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1281162
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia, Overweight, Cardiovascular Risk, Obesity
MeSH Terms: conditions — Schizophrenia; Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 500 patients: Patients with diagnosis of schizophrenia, schizophreniform or schizoaffective disorder (DSM-IV TR) with BMI (body mass index) more or equal to 25 Kg/m2
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — non-interventional

SUMMARY:
To analyse the progress of modifiable metabolic risk factors (Blood pressure, cigarette smoking, waist perimeter, BMI, glycemia and lipidic profile) in schizophrenic patients with overweight for 12 months.

To analyse the perceived health status and the level of functioning and disability of patients with schizophrenia and overweight and their progress at 3, 6 and 12 months.

To assess the progress of the symptoms of the disease at 6 and 12 months.

DETAILED DESCRIPTION:
Consecutive patient sampling. Any investigational site four consecutive patients with diagnosis of Schizophrenia (DSM-IV TR) and Overweight (BMI more or equal to 25 Kg/m2)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of schizophrenia, schizophreniform or schizoaffective disorder (DSM-IV TR)
* Patients with BMI (body mass index) more or equal to 25 Kg/m2
* Patients or their legal representative have provided written informed consent

Exclusion Criteria:

* Patients are unable to complete or to understand health questionnaires in Spanish language
* Patients are currently enrolled on clinical trials or other investigational studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample. Patients >17 years older with diagnosis of Schizophrenia (DSM-IV TR) and Overweight (BMI more or equal to 25 Kg/m2)
Sampling Method: Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evolution of modifiable metabolic risk factors (Blood pressure, cigarette smoking, waist perimeter, BMI, glycemia and lipidic profile) in schizophrenic patients with overweight for 12 months. | 12 months

SECONDARY OUTCOMES:
Cardiovascular Risk | 12 months
To assess the progress of the symptoms and clinical evolution of the disease | 12 months
Patient Functional Impairment | 12 months
Patient Quality of Life | 12 months
Current Pattern of Treatment in this Population | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281162&StudyName=Control%20of%20Metabolic%20and%20Cardiovascular%20Risk%20in%20Patients%20with%20Schizophrenia%20and%20Overweight